CLINICAL TRIAL: NCT02701049
Title: Emergency Department Query For Patient-centered Approaches To Sexual Orientation And Gender Identity
Brief Title: Patient Centered Methods to Collect Sexual Orientation and Gender Identity Status in the ED
Acronym: EQUALITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Adil Haider, Kessler Director, Center for Surgery and Public Health, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015P002475
Record Dates: First submitted 2016-01-07; First posted 2016-03-08 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Homosexuality; Gender Identity
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SO/GI Collection (Other): Methods to collect SO/GI information in the ED
  Interventions: Other: Methods to collect SO/GI information in the ED

INTERVENTIONS:
Other: Methods to collect SO/GI information in the ED — In Mode 1, all patients presenting to the ED will have SO/GI information collected verbally by the nurse, which is standard of care. In Mode 2, all patients presenting to the ED will have SO/GI information collected in a non-verbal manner, in which the registrar will ask them to complete an electronic form.

SUMMARY:
This trial is the final phase of a three phase PCORI-funded study to develop and test patient-centered approaches to collect sexual orientation and gender identity (SO/GI) information in the ED. From the results of Phase 1 qualitative interviews and national quantitative survey and Phase 2 Delphi rounds with the Stakeholder Advisory Board, we have determined two methods of collection favored by patients and providers to implement in the trial. The first method, nurse verbal collection, is in alignment with Partners recommended clinical practice and is therefore a quality improvement (QI) evaluation. The second method, non-verbal registrar form collection with nurse verbal confirmation, is a research intervention to evaluate and compare a new patient-centered approach to SO/GI collection. To compare the patient-centeredness of the two different approaches, satisfaction surveys will be administered to ED patients and staff members involved in collection.

In summary, the study design (1) evaluates recommended current practice (QI), (2) evaluates a quality improvement project to increase recommended current practice, and (3) evaluates a new method of collecting SO/GI (research intervention).

ELIGIBILITY:
Inclusion Criteria:

* Adult ED patients who are cognitively and physically capable of informed consent
* Adult ED nurses and registrars who are cognitively and physically capable of informed consent

Exclusion Criteria:

* Children
* Any person not cognitively and physically capable of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Haider, MD, MPH, Principal Investigator — Brigham and Women's Hospital

REFERENCES:
- [Background] De Santis JP. HIV infection risk factors among male-to-female transgender persons: a review of the literature. J Assoc Nurses AIDS Care. 2009 Sep-Oct;20(5):362-72. doi: 10.1016/j.jana.2009.06.005. PMID 19732695
- [Background] Lombardi EL, Wilchins RA, Priesing D, Malouf D. Gender violence: transgender experiences with violence and discrimination. J Homosex. 2001;42(1):89-101. doi: 10.1300/j082v42n01_05. PMID 11991568
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: HIV testing and diagnosis among adults--United States, 2001-2009. MMWR Morb Mortal Wkly Rep. 2010 Dec 3;59(47):1550-5. PMID 21124295
- [Background] Struble CB, Lindley LL, Montgomery K, Hardin J, Burcin M. Overweight and obesity in lesbian and bisexual college women. J Am Coll Health. 2010;59(1):51-6. doi: 10.1080/07448481.2010.483703. PMID 20670929
- [Background] Buchmueller T, Carpenter CS. Disparities in health insurance coverage, access, and outcomes for individuals in same-sex versus different-sex relationships, 2000-2007. Am J Public Health. 2010 Mar;100(3):489-95. doi: 10.2105/AJPH.2009.160804. Epub 2010 Jan 14. PMID 20075319
- [Background] Dilley JA, Simmons KW, Boysun MJ, Pizacani BA, Stark MJ. Demonstrating the importance and feasibility of including sexual orientation in public health surveys: health disparities in the Pacific Northwest. Am J Public Health. 2010 Mar;100(3):460-7. doi: 10.2105/AJPH.2007.130336. Epub 2009 Aug 20. PMID 19696397
- [Background] Herbst JH, Jacobs ED, Finlayson TJ, McKleroy VS, Neumann MS, Crepaz N; HIV/AIDS Prevention Research Synthesis Team. Estimating HIV prevalence and risk behaviors of transgender persons in the United States: a systematic review. AIDS Behav. 2008 Jan;12(1):1-17. doi: 10.1007/s10461-007-9299-3. Epub 2007 Aug 13. PMID 17694429
- [Background] Whitbeck LB, Chen X, Hoyt DR, Tyler KA, Johnson KD. Mental disorder, subsistence strategies, and victimization among gay, lesbian, and bisexual homeless and runaway adolescents. J Sex Res. 2004 Nov;41(4):329-42. doi: 10.1080/00224490409552240. PMID 15765273
- [Background] Diaz RM, Ayala G, Bein E, Henne J, Marin BV. The impact of homophobia, poverty, and racism on the mental health of gay and bisexual Latino men: findings from 3 US cities. Am J Public Health. 2001 Jun;91(6):927-32. doi: 10.2105/ajph.91.6.927. PMID 11392936

RESULTS

PARTICIPANT FLOW:
Groups:
- Mode 0: Patients who were not asked their SO/GI
- Mode 1: Patients who were verbally asked by a nurse their SO/GI
- Mode 2: Patients whose SO/GI was collected non-verbally on a form
Period: Overall Study
Arm/Group | Mode 0 | Mode 1 | Mode 2
Started | 209 (Patients who completed a follow-up survey) | 342 (Patients who completed a follow-up survey) | 198 (Patients who completed a follow-up survey)
Completed | 209 (Total patients included in analysis) | 342 (Total patients included in analysis) | 198 (Total patients included in analysis)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients who were not asked their SO/GI or who provided their SO/GI in the ED via verbal or nonverbal collection and completed a patient outcome survey
Groups:
- Total: Total of all reporting groups
Arm/Group | Mode 0 | Mode 1 | Mode 2 | Total
Number analyzed (Participants) | 209 | 342 | 198 | 749
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 48 (17.2) | 38.5 (13.5) | 33 (12.3) | 39.3 (15.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 97 | 75 | 32 | 204
  Female | 107 | 149 | 85 | 341
  Transgender Male to Female | 0 | 1 | 1 | 2
  Transgender Female to Male | 0 | 3 | 2 | 5
  Queer/Genderqueer | 0 | 0 | 1 | 1
  Questioning/Unsure | 0 | 0 | 1 | 1
  Declined to State | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0
  Unavailable/Not Asked | 5 | 114 | 74 | 193
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 69 | 123 | 77 | 269
  Black | 78 | 178 | 85 | 341
  Asian | 4 | 3 | 2 | 9
  American Indian | 0 | 1 | 3 | 4
  Native Hawaiian | 0 | 0 | 1 | 1
  Hispanic | 17 | 30 | 25 | 72
  Other | 3 | 4 | 4 | 11
  Unknown | 3 | 2 | 0 | 5
  Declined | 1 | 1 | 1 | 3
  Missing | 34 | 0 | 0 | 34

OUTCOME MEASURES:

1. Primary Outcome: Communication Climate Assessment Toolkit Questionnaire (Patient)
Description: The primary outcome was patient satisfaction as measured by a modified Communication Climate Assessment Toolkit (CCAT) patient survey, an assessment of attitudes towards organizational climate and provider/patient communication.The CCAT is reliable, validated in geographically and ethnically diverse health care organizations, and accurately predicts patient-reported quality and trust. Containing 5/7 items from the full CCAT, our pre-specified modified scale included only questions that were applicable to the ED population, e.g. we kept the question "Do you feel welcome at the hospital?" but eliminated the question "Was it easy to reach someone on the phone if you had a question?" from analyses.Each scale item was scored as a 0 (most disagreement), ½ (neutral), or 1 (agreement), resulting in a scale score ranging from 0-5; higher scores were considered more favorable. The average score for the modified scale was calculated and multiplied by 20 to provide the overall score out of 100.
Time Frame: Through study completion (approximately 1 year)
Population: Patients who were not asked SO/GI or who provided their SO/GI in the ED via verbal or nonverbal collection and provided complete data on the patient outcome survey
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Mode 0 | Mode 1 | Mode 2
Number analyzed (Participants) | 209 | 342 | 198
Score | 92.78 (18.05) | 91.32 (18.52) | 94.14 (13.44)

2. Secondary Outcome: Staff-reported Outcomes Measure Questionnaire
Description: Measures responses to the staff survey question, "Did you experience difficulty collecting sexual orientation data from patients?"
Time Frame: Through study completion (approximately 1 year)
Population: Nurses and registrars who completed staff outcome surveys
Measure: Count of Participants; unit: Participants
Groups:
- Mode 1: Nurses who verbally collected SO/GI
- Mode 2: Registrars who collected SO/GI non-verbally on a form
Arm/Group | Mode 1 | Mode 2
Number analyzed (Participants) | 41 | 38
Participants
  Never/rarely | 11 | 14
  Sometimes | 16 | 14
  Usually/Always | 7 | 8
  Other | 6 | 2
  Decline to answer | 1 | 0

3. Secondary Outcome: Proportion of Patients Reporting SO/GI
Description: Measures the proportion of all adult emergency department patients from whom SO/GI was collected during the study period
Time Frame: Through study completion (approximately 1 year)
Population: All adult patients who were seen in the ED during the intervention periods
Measure: Count of Participants; unit: Participants
Groups:
- Mode 1; Mode 2: Patients who had SO/GI recorded in the EHR of all adult ED patients
Arm/Group | Mode 1 | Mode 2
Number analyzed (Participants) | 342 | 198
Participants | 228 | 132
Statistical Analysis 1: Comparison: Mode 1 vs Mode 2; Historical controls included all patients entering participating EDs as identified by the Electronic Health Record; Test type: Other — Among 109,994 patients who entered the ED during Mode 1, 19,742 had SOGI collected (18%). Among 88,143 patients who entered the ED during Mode 2, 3,630 had SOGI collected (4%); Results were compared to historical control population from an electronic health record database, no other data were collected for these participants

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Mode 0 | Mode 1 | Mode 2
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/342 | 0/198
Serious Adverse Events (participants affected / at risk) | 0/209 | 0/342 | 0/198
Other Adverse Events (participants affected / at risk) | 0/209 | 0/342 | 0/198

LIMITATIONS AND CAVEATS:
Patients who identified their SO/GI as "other" were not eligible for inclusion in the study. Patients who were admitted to the ED with a psychiatric diagnosis were not eligible for participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT02701049/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT02701049/Prot_SAP_001.pdf